CLINICAL TRIAL: NCT04546191
Title: Symptoms and Wellbeing of People Infected With Covid-19 Virus in Iceland
Status: Completed | Type: Observational
Sponsor: Landspitali University Hospital (Other)
Responsible Party: Principal Investigator, Helga Jónsdóttir, Professor, Landspitali University Hospital
Other Study IDs: LSH-20-002
Record Dates: First submitted 2020-09-10; First posted 2020-09-11 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Covid19
Keywords: Covid19; Symptoms; Well being; Survey
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this cross-sectional study is to explore symptoms and well being of people diagnosed with COVID-19 from the outset of the pandemic until June 2020.

DETAILED DESCRIPTION:
All patients diagnosed with COVID-19 in Iceland were referred to the COVID-19 outpatient clinic at Landspitali National University Hospital in Iceland. In the clinic risk assessment was conducted and the patients were accordingly provided with individualized care be it telephone surveillance, onsite examination and treatment, or admission to the hospital. As the the first wave of the pandemic was curbing the necessity of exploring how the patients did and continue to fare after being infected became apparent.

The research questions are:

What were the symptoms that patients expressed during and about three months after being diagnosed with COVID-19? What is the prevalence and intensity of the symptoms that patients expressed during and about three months after being diagnosed with COVID-19 ? How do patients value their health related quality of life, what is their health literacy and sense of security in care during and about three months after being diagnosed with COVID-19 ? How do patients value the nursing care in the outpatient COVID-19 clinic? What are the patients' perception of having caught COVID-19?

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving care from the COVID-19 outpatient clinic at LUH during the first wave of the pandemic

Exclusion Criteria:

* Young than 18 y.o.
* Do not understand Icelandic
* Died

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients receiving care from the COVID-19 outpatient clinic at LUH during the first wave of the pandemic
Sampling Method: Non-Probability Sample
Enrollment: 1580 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Symptoms | 2 months
  Patients answer a questionnaire developed by authors based on published symptoms of COPVID19. The questionnare has two versions one refers to symptoms during the quarantine and the other to the time a couple of months later. Name: Symptoms during and after the COVID 19 quarantine.
  The questionnaire has 25 items scored on a four point Likert scale. The highest possible score is 100 and the lowest possible score is 20. Higher score means worse outcome.

SECONDARY OUTCOMES:
Wellbeing - HRQL | 2 months
  EQ-5D is a generic health related quality of life measurement (HRQL). It is composed of five dimensions; mobility, self-care, usual activities, pain/discomfort and anxiety/depression measured on five levels (from no problems to extreme problems or unable) with a minimum score 5 and maximum score 25, with higher score indicating worse outcome. The instrument contains as well a visual analogue scale (VAS) measuring the person's "health state today", on a 100 point scale (worst imaginable to best imaginable health state).

OTHER OUTCOMES:
Anxiety and depression (HADS) | 2 months
  Hospital Anxiety and Depression Scale (HADS) is a widely used instrument to assess anxiety and depression in people attending outpatient hospital clinics. Sensitive to mild disturbances, HADS is a reliable and valid instrument consisting of a 14 item 4 point (0-3) Likert scale with two subscales; anxiety (7 items) and depression (7 items). The minimum score is 0 and the highest possible score is 42. Higher score refers to worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Brynja Ingadottir, PhD, Principal Investigator — Faculty of Nursing
Locations (1):
- Landspitali National University Hospital, Reykjavik, Ísland, Iceland